CLINICAL TRIAL: NCT07028840
Title: A Comparison of Extracorporeal Shockwave Therapy (ESWT) and High-intensity Laser Therapy (HILT) in Terms of Pain, Function and Grip Strength in Lateral Epicondilitis: a Randomized Controlled Study
Brief Title: Physiotherapy Applications in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Suat EREL, HEAD OF THE DEPARTMENT OF ORTHOPEDIC REHABILITATION, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 674325
Record Dates: First submitted 2021-10-07; First posted 2025-06-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Physical Therapy Modalities; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physiotherapy (Active Comparator): This group received conventional physiotherapy only
  Interventions: Other: Physiotherapy
- Physiotherapy + ESWT (Active Comparator): This group received conventional physiotherapy and additional extracorporeal shock wave therapy (ESWT)
  Interventions: Other: Physiotherapy; Device: Extracorporeal Shock Wave Therapy (ESWT)
- Physiotherapy + HILT (Active Comparator): This group received conventional physiotherapy and additional high-intensity laser therapy (HILT).
  Interventions: Other: Physiotherapy; Device: High-Intensity Laser Therapy (HILT)

INTERVENTIONS:
Other: Physiotherapy — 10 sessions over 2 weeks, including TENS, cold therapy, ultrasound, and exercise therapy, 5 sessions per week.
Device: Extracorporeal Shock Wave Therapy (ESWT) — 4 sessions total, applied 2 times per week for 2 weeks.
  Arms: Physiotherapy + ESWT
Device: High-Intensity Laser Therapy (HILT) — 4 sessions total, applied 2 times per week for 2 weeks.
  Arms: Physiotherapy + HILT

SUMMARY:
This study aims to compare the effectiveness of extracorporeal shock wave therapy (ESWT) and high-intensity laser therapy (HILT) in improving pain, grip strength, and function in patients with lateral epicondylitis. A total of 42 volunteer patients aged 18-65 were enrolled at Balıkesir Private Sevgi Hospital physical medicine polyclinic. Participants were randomly assigned into three groups: group 1 received conventional physiotherapy, group 2 received physiotherapy plus ESWT, and group 3 received physiotherapy plus HILT. Physiotherapy was applied for 2 weeks, totaling 10 sessions. ESWT and HILT were each administered twice weekly for 2 weeks, totaling 4 sessions. Pain was measured using the visual analog scale (VAS), grip strength with a hand dynamometer, and function using the Duruöz Hand Index and PRTEE-T questionnaire. Evaluations were performed before treatment, after 2 weeks, and one month post-treatment.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the effects of extracorporeal shock wave therapy (ESWT) and high-intensity laser therapy (HILT) on pain, grip strength, and function in patients diagnosed with lateral epicondylitis. The study was conducted at the physical medicine polyclinic of Balıkesir Private Sevgi Hospital and included 42 patients aged 18 to 65 who were referred for therapeutic physical therapy after being diagnosed for the first time with lateral epicondylitis.

Participants were randomly divided into three groups:

Group 1: received conventional physiotherapy including hot pack application, transcutaneous electric nerve stimulation (TENS), and stretching/strengthening exercises. Physiotherapy was administered 5 times per week for 2 weeks (total of 10 sessions).

Group 2: received the same physiotherapy as group 1, plus extracorporeal shock wave therapy (ESWT) administered twice per week for 2 weeks (total of 4 sessions).

Group 3: received the same physiotherapy as group 1, plus high-intensity laser therapy (HILT) administered twice per week for 2 weeks (total of 4 sessions).

Pain severity was evaluated using the visual analog scale (VAS), grip strength using a hand dynamometer, and functional status using the Duruöz Hand Index and patient-rated tennis elbow evaluation (PRTEE-T). All outcome measures were assessed at three time points: baseline (before treatment), post-treatment (after 2 weeks), and at 1-month follow-up. The primary objective was to assess whether either ESWT or HILT offers additional benefit over standard physiotherapy and whether one modality is superior to the other in treating lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18,
* Being diagnosed with lateral epicondylitis,
* Not having received lateral epicondylitis treatment in the last 3 months

Exclusion Criteria:

* Stopping the treatment,
* Those who have been traumatized in the last 3 months,
* Those who use drugs that can affect muscle strength or pain level (muscle relaxants, analgesics, gabapentinoids, etc.)
* Those with open wounds in the elbow area, Those with elbow fractures, Those with drug allergies, Pregnant and breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Pain Severity - Visual Analog Scale (VAS) | Baseline (Day 1), at the end of 2-week treatment, 4 weeks after treatment completion
  Pain intensity will be evaluated using the visual analog scale (VAS), a 10 cm line ranging from 0 (no pain) to 10 (worst imaginable pain). Continuous scale (0-10), higher scores indicate worse outcome.
Grip Strength - Hand Dynamometer | Baseline (Day 1), at the end of 2-week treatment, 4 weeks after treatment completion
  Grip strength will be measured in kilograms using a hand dynamometer. Continuous scale, higher scores indicate better outcome
Upper Extremity Function - Duruöz Hand Index | Baseline (Day 1), at the end of 2-week treatment, 4 weeks after treatment completion
  The Duruöz Hand Index is a functional scale that assesses hand-related disability. Scores range from 0 to 90, with higher scores indicating worse functional impairment.
Functional Evaluation - PRTEE-T (Patient-Rated Tennis Elbow Evaluation) | Baseline (Day 1), at the end of 2-week treatment, 4 weeks after treatment completion
  The PRTEE-T is a 15-item patient-rated questionnaire for lateral epicondylitis. Total scores range from 0 (no disability) to 100 (maximum disability). Continuous scale (0-100), higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: SUAT EREL, PROF.DR., Study Director — PAMUKKALE UNİVERSİTY
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: FOR 6 MONTH
Access Criteria: FOR RESEARCH